CLINICAL TRIAL: NCT01486537
Title: Characterization of Blood Drawn From the Pulp of Primary Molar Undergoing Pulpotomy or Pulpectomy.
Brief Title: Acidity Level of Blood From Primary Molar's Pulp While Undergoing Pulpotomy or Pulpectomy Procedure
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moti Moskovitz, dr, Hadassah Medical Organization
Other Study IDs: pulpastrop-HMO-CTIL
Record Dates: First submitted 2011-12-03; First posted 2011-12-06 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Healthy
Keywords: samples; children; the age group 3-13 years

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood specimens which are undergoing Astrop test (acidity level .po2 pco2)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- theeth undergoing pulpotomy
- teeth undergoing pulpectomy

SUMMARY:
The aim of this study is to evaluate the level of acidity of blood samples that are been taken from pulp chambers of primary molars undergoing pulpotomy or pulpectomy procedures. Our hypothesis is that samples from teeth undergoing pulpectomy would be acidic while samples from teeth undergoing pulpotomy would bo neutral.

DETAILED DESCRIPTION:
The samples will be collected by 1 m"l syringe that is pre-washed with Heparin.than the samples will be analyzed in an Astrop machine of neonates.

ELIGIBILITY:
Inclusion Criteria:

* no systemic disease
* teeth that are undergoing pulpotomy or pulpectomy

Exclusion Criteria:

* systemic disease
* pulp necrosis
* permanent teeth

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children undergoing dental treatment by residents in Hadassah hospital Jerusalem.
  Ages between 3-13 years old.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2011-12; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moti Moskovitz, Dr., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel